CLINICAL TRIAL: NCT00678444
Title: Patient Satisfaction Regarding Timing of Clean Intermittent Self-Catheterization Teaching After Prolapse or Incontinence Surgery
Brief Title: Patient Satisfaction Study: Clean Intermittent Self-Catheterization Teaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PRO07070018
Record Dates: First submitted 2008-05-10; First posted 2008-05-15 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2016-10

CONDITIONS: Anxiety
Keywords: Anxiety; Satisfaction; Incomplete bladder emptying; Clean Intermittent Self-catheterization; Prolapse/incontinence surgery
MeSH Terms: conditions — Anxiety Disorders; Personal Satisfaction; Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Non-educational video self-cath (No Intervention): Randomized to not watching educational video about clean intermittent self-catheterization prior to prolapse/incontinence surgery.
- Arm 2: Educational Video Self-cath (Experimental): Randomized to watch educational video about clean intermittent self-catheterization prior to prolapse/incontinence surgery.
  Interventions: Other: Educational video

INTERVENTIONS:
Other: Educational video — Watching an educational video about clean intermittent self-catheterization prior to prolapse/incontinence surgery.
  Arms: Arm 2: Educational Video Self-cath

SUMMARY:
To compare patient satisfaction and anxiety scores between female subjects undergoing urinary incontinence and/or pelvic reconstructive surgery who are instructed preoperatively in the technique of clean intermittent self-catheterization (CISC) by means of an instructional video and those who do not receive specific preoperative instruction in CISC, other than basic informed consent regarding risks of postoperative urinary retention.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment will be offered to all women undergoing pelvic reconstructive and/or urinary incontinence surgery by the DIvision of Urogynecology, Department of Obstetrics and Gynecology at Magee Womens Hospital.

Exclusion Criteria:

* Subjects who have performed CISC in the past will be excluded.
* Subjects whose score on the MMSE reflects dementia (<24) will be excluded.
* Subjects anticipated to have placement of a suprapubic catheter placement at the time of surgery will be excluded.
* Subjects deemed by the enrolling physician to be incapable of physically performing self-catheterization will be excluded.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2008-04; Primary Completion 2011-04 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry L Lowder, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center - Center for Female Bladder and Pelvic Health, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Non-educational Video Self-catheterization: Patients in this group will not watch the educational video about clean intermittent self-catheterization prior to prolapse/incontinence surgery
- Arm 2: Educational Video Self-catheterization Group: Randomized to watch pre-operative educational video about clean intermittent self-catheterization prior to prolapse/incontinence surgery.
Period: Overall Study
Arm/Group | Arm 1: Non-educational Video Self-catheterization | Arm 2: Educational Video Self-catheterization Group
Started | 100 | 99
Completed | 100 | 99
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomized to Not Watch Educational Video: Randomized to not watch pre-operative educational video about clean intermittent self-catheterization prior to prolapse/incontinence surgery.
- Randomized to Watch Pre-operative Educational Video About Clea: Randomized to watch pre-operative educational video about clean intermittent self-catheterization prior to prolapse/incontinence surgery.
- Total: Total of all reporting groups
Arm/Group | Randomized to Not Watch Educational Video | Randomized to Watch Pre-operative Educational Video About Clea | Total
Number analyzed (Participants) | 100 | 99 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (9.8) | 59.7 (11.7) | 58.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 99 | 199
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 99 | 95 | 194
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 100 | 99 | 199
Mini-Mental Status Examination [Median (Inter-Quartile Range); unit: units on a scale] — Range: 0-30. Higher score represents better cognitive function.
  units on a scale | 30 [29 to 30] | 30 [29 to 30] | 30 [29 to 30]
Pelvic Floor Distress Inventory-20 [Median (Inter-Quartile Range); unit: units on a scale] — Range: 0-300 (total) Higher score represents more bother from pelvic floor disorder symptoms.
  units on a scale | 84 [56 to 120] | 103 [64 to 142] | 94 [60 to 131]
Pelvic Floor Impact Questionnaire-7 [Median (Inter-Quartile Range); unit: units on a scale] — Range: 0-300 Higher score represents greater impact of pelvic floor disorders on quality of life.
  units on a scale | 41 [19 to 93] | 59 [33 to 105] | 50 [26 to 99]
Personal Health Questionnaire-9 [Median (Inter-Quartile Range); unit: units on a scale] — Range: 1-27 Higher scores represent worsening degrees of depression.
  units on a scale | 2 [0 to 5] | 2 [0 to 5] | 2 [0 to 5]
State-Trait Anxiety Inventory-State scale [Mean (Standard Deviation); unit: units on a scale] — Range: 40-160. Higher score represents higher anxiety level/more anxiety.
  units on a scale | 37.9 (11.6) | 40.7 (11.7) | 39.3 (11.7)

OUTCOME MEASURES:

1. Primary Outcome: State-Trait Anxiety Inventory-State Scores
Description: The STAI-S scale is a 20-item, Likert-type, validated measure, scored 20-80 with higher scores reflecting higher situational anxiety. STAI-S is designed to specifically assess current anxiety as opposed to baseline trait anxiety. Respondents rated their current feelings specific to bladder catheterization by answering items regarding bladder catheterization such as, "I feel at ease" or "I feel upset." Responses ranged from 1 to 5 from "not at all" to "very much so."
Time Frame: Baseline, after viewing educational video, after learning self-cathterization, 6 weeks post-operatively
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: Education Without Video Tutorial: Patients in this group will not watch the educational video about clean intermittent self-catheterization prior to prolapse/incontinence surgery
- Randomized to Watch Educational Video About Clean Intermittent: Randomized to watch educational video about clean intermittent self-catheterization prior to prolapse/incontinence surgery.
Arm/Group | Arm 1: Education Without Video Tutorial | Randomized to Watch Educational Video About Clean Intermittent
Number analyzed (Participants) | 100 | 99
units on a scale
  Baseline | 37.9 (11.6) | 40.7 (11.7)
  Post-video | NA (NA) — Not measured as this group did not view video at this time point. | 37.7 (12.5)
  Voiding Trial Failure | 40.6 (9.7) | 42.5 (11.9)
  Discharge | 33.4 (11.7) | 35.6 (13.0)
  6-weeks postoperative | 30.2 (10.9) | 32.7 (13.4)

2. Secondary Outcome: Patient Satisfaction Scores - Visual Analogue Scores (VAS).
Description: Secondary study measures included a study-specific visual analog scales (VAS, range 0-100 mm) to assess comfort with Clean Intermittent Self-Catheterization (CISC) and opinions on the CISC video.
  Higher VAS scores represent higher levels of comfort with CISC.
Time Frame: Baseline, post-operatively at time of discharge from hospital, 6 weeks post-operatively
Measure: Number; unit: participants
Arm/Group | Arm 1: Education Without Video Tutorial | Randomized to Watch Educational Video About Clean Intermittent
Number analyzed (Participants) | 100 | 99
participants
  Baseline-Comfort level | 36 | 36
  Baseline-Worry | 44 | 44
  Baseline-CISC affect Satisfaction | 7 | 7
  Baseline-Feels catheterization would be difficult | NA — Routine care group did not view video. | 32
  After viewing video-Video Helpful | NA — Routine care group did not view video. | 95
  After viewing video-Worry | NA — Routine care group did not view video. | 31
  After viewing video-Relieving fear/anxiety | NA — Routine care group did not view video. | 82
  After viewing video-Comfort with catheterization | NA — Routine care group did not view video. | 52
  Postvideo-Feels catheterization would be difficult | NA — Routine care group did not view video. | 22

ADVERSE EVENTS:
Time Frame: Adverse events were reported for the 8-week period of the study starting with the pre-operative visit where participants wre randomized to the Video versus usual treatment arm.
Groups:
- Arm 1: Non-educational Video Self-catheterization Group: Patients in this group will not watch the educational video about clean intermittent self-catheterization prior to prolapse/incontinence surgery
- Arm 2: Educational Video Self-catheterization Group: Randomized to watch educational video about clean intermittent self-catheterization prior to prolapse/incontinence surgery.
Arm/Group | Arm 1: Non-educational Video Self-catheterization Group | Arm 2: Educational Video Self-catheterization Group
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/99
Other Adverse Events (participants affected / at risk) | 34/93 | 32/91
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Non-educational Video Self-catheterization Group (N=93) | Arm 2: Educational Video Self-catheterization Group (N=91)
Failed post-operative voiding trial (Renal and urinary disorders) | 34 (34) | 32 (32) — Failed post-operative voiding trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No